CLINICAL TRIAL: NCT00521495
Title: Carpal Tunnel Syndrome and Static Magnetic Field Therapy
Acronym: CTS/SMF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Natural Medicine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Oregon Health and Science University (Other)
Responsible Party: Agatha Colbert, Principal Investigator, National College of Natural Medicine
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R21AT003293 (NIH); R21AT003293 (NIH)
Record Dates: First submitted 2007-08-24; First posted 2007-08-28 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Carpal Tunnel Syndrome
Keywords: static magnetic field; permanent magnet; carpal tunnel syndrome; median nerve
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Surface magnetic field strength at target 450 Gauss permanent magnet
  Interventions: Device: neodymium permanent magnet; Device: neodymium magnet
- B (Experimental): Surface field strength at target 150 Gauss permanent magnet
  Interventions: Device: neodymium magnet
- C (Active Comparator)
  Interventions: Device: neodymium magnet; Device: magnet

INTERVENTIONS:
Device: neodymium permanent magnet — 3/4" diameter by 1/8" thick permanent magnet
  Arms: A
Device: neodymium magnet — A. 450 Gauss static magnetic field at target B. 150 Gauss static magnetic field at target C. 0 Gauss static magnetic field at target
Device: magnet — 0 Gauss magnets are worn every night during hours of sleep for 6 weeks.
  Arms: C

SUMMARY:
The purpose of this Phase II study is to assess the feasibility of conducting a large scale trial which will evaluate the effectiveness of static magnetic field therapy as a treatment for Carpal Tunnel Syndrome. This preliminary study will determine which of three strength magnets to use in the future.

Participants will be recruited from three primary sources. 1) Patients with a possible diagnosis of Carpal Tunnel Syndrome who have been referred to the Orthopaedic and Rehabilitation Clinics of OHSU for Nerve conduction studies. If after conducting these studies a potential participant shows evidence of mild to moderate Carpal Tunnel Syndrome s/he will be informed about the study and invited to participate in additional screening. B) Patients seen at the National College of Natural Medicine (NCNM) Clinics who have a clinical diagnosis of Carpal Tunnel Syndrome will be informed about the study and invited to enter the screening process for further eligibility. C) Participants will also be recruited from the general public including staff and students at OHSU and NCNM).

Eligibility will be determined through a stepwise process including telephone screening for general eligibility, Nerve Conduction screening for electrodiagnostic eligibility, and Boston Carpal Tunnel Questionnaire screening for symptom severity eligibility. Those potential participants who meet all eligibility requirements will be randomized to one of three magnetic field dosages. They will be provided with a ¾" diameter x 1/8" thick magnet which they will be required to apply for six weeks during the hours of sleep. Over the course of the study participants will have four visits to the General Clinical Research Center of OHSU and three visits to the Orthopaedic and Rehabilitation Clinics of OHSU for Nerve Conduction studies to be performed by either Dr. Nels Carlson or Dr. Hans Carlson.

Questionnaires to be completed during the course of the study include a general health information and demographics questionnaire, the Boston Carpal Tunnel Questionnaire, which will be completed on six occasions, a general symptoms checklist and a Post Treatment Participant satisfaction questionnaire.

Recruitment, retention, compliance and safety will be analyzed using descriptive statistics. Effectiveness of the three different strength magnets will be assessed by comparing participants' baseline scores on the Boston Carpal Tunnel Questionnaire with their scores after six weeks of magnet use.

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion Criteria:

Age range (18-65 years) Both genders Hand or wrist pain with paresthesias or numbness in any or all fingers, predominating in a median nerve distribution, and especially occurring at night Symptoms present for at least 3 months No prior treatment with magnet therapy Baseline BCTQ >2.0 on SSS subscale Meet specific EDX inclusion/ exclusion criteria listed in Table 1 (below) Willing and able to provide informed consent Ability to read English fluently

Exclusion Criteria:

Use of narcotic analgesia Corticosteroid injection into the carpal tunnel within previous 3 months Prior carpal tunnel surgery on affected side History of wrist or hand fracture on the symptomatic limb Skin rash or irritation on the wrist Participant (or bed partner) wearing a pacemaker or other electronic device Current pregnancy, less than 3 months postpartum, nursing, or planning a pregnancy Plans to move from area during the time frame of the study Inability to tolerate the baseline screening nerve conduction study Unable or unwilling to comply with the protocol Collecting workers' compensation or social-security disability benefits Involved in litigation regarding pain or disability Development of a rash or skin irritation to the tape applied to the wrist during a run-in baseline test period

Concomitant medical conditions including:

Insulin-dependent diabetes mellitus History of chronic renal failure or renal dialysis or forearm fistulae History of generalized peripheral neuropathy History of other neurologic disorders which may confuse the diagnosis of carpal tunnel syndrome, including but not limited to stroke, cervical radiculopathy, myelopathy, subdural hematoma, brain tumor Inflammatory articular disease or tendonitis of the involved hand or wrist Other disorders known to predispose to carpal tunnel syndrome including acromegaly, multiple myeloma, amyloidosis Cancer

Table 1. Electrodiagnostic (EDX) Inclusion and Exclusion Criteria Inclusion Criteria

* Median nerve onset sensory latency > 3.5 ms at 13 cm
* Median-ulnar across palm latency difference ≥ 0.4 ms
* Median-radial to thumb latency difference ≥ 0.7 ms
* Median-ulnar to ring finger latency difference ≥ 0.5ms ED Exclusion Criteria
* Absent sensory nerve action potential (SNAP)
* Median nerve distal motor latency > 6.0 ms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-06 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Questionnaire Symptom Severity Scale | Baseline, Wks 2, 4, 6, 18

SECONDARY OUTCOMES:
1. Electrophysiological recovery of median nerve | Baseline, 6 weeks, 18 weeks
2. General symptom questionnaire | Baseline and on completion of intervention phase
3. Compliance with treatment | Baseline to study completion

CONTACTS AND LOCATIONS:
Overall Officials: Agatha P Colbert, MD, Principal Investigator — National University of Natural Medicine
Locations (1):
- National College of Natural Medicine, Portland, Oregon, United States

REFERENCES:
- [Derived] Colbert AP, Markov MS, Carlson N, Gregory WL, Carlson H, Elmer PJ. Static magnetic field therapy for carpal tunnel syndrome: a feasibility study. Arch Phys Med Rehabil. 2010 Jul;91(7):1098-104. doi: 10.1016/j.apmr.2010.02.013. PMID 20599049